CLINICAL TRIAL: NCT02423681
Title: Evaluation of Overall Therapy Cost Comparing First Intention and Second Intention Heated Humidification for CPAP: A Pilot Study.
Brief Title: A Comparison of CPAP With and Without Humidification: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CIA-101
Record Dates: First submitted 2015-04-15; First posted 2015-04-22 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Heated humidification as first intention (HH1st) (Active Comparator): Subjects receive heated humidification as first intention with ThermoSmart
  Interventions: Device: ThermoSmart
- Non-heated humidification (Placebo Comparator): Subjects will receive no humidification. However they can be switched to the humidification group if patients complains of nasal dryness, congestion, nose bleed or if they had significant leak that cannot be resolved by two changes of mask.
  Interventions: Device: Without ThermoSmart

INTERVENTIONS:
Device: ThermoSmart — Heated humidification as first intention (HH1st) with ThermoSmart
  Arms: Heated humidification as first intention (HH1st)
Device: Without ThermoSmart — ThermoSmart is switched off
  Arms: Non-heated humidification

SUMMARY:
To compare a group of patients with our standard treatment of continuous positive airway pressure (CPAP) and another group of patients with CPAP and a humidifier attached. The therapy cost and the successfulness of the treatment will be measured. A humidifier is a water chamber that is currently added to CPAP only if the patients needs it.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years of age
* Diagnosed with OSA (obstructive sleep apnea) and eligible for CPAP treatment under local requirements (NICE guidelines: AHI (apnea hypopnea index) ≥ 15, or AHI > 5 with significant daytime sleepiness)
* Naïve to CPAP therapy, i.e. have not been prescribed, or used CPAP in the last 5 years.
* Fluent in spoken and written English

Exclusion Criteria:

* Significant uncontrolled cardiac disease, as per the principal investigator's discretion
* Co-existing lung disease, as per the principal investigator's discretion
* Co-existing sleep disorder, such a predominant central sleep apnoea
* Pregnancy
* Participants that are unable or unwilling to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Overall cost of equipment | 6 months
  (cost of equipment required for CPAP therapy, including CPAP device and mask, and all related consumables
Number and type of additional interventions | 6 months
  The number and type of additional interventions (masks, nasal steroids) and the associated cost
Duration of appointments | 6 months
  Time spent with/on each patient (i.e preparation and follow-up time as well as appointment time)
Number of unplanned follow-ups | 6 months
  number of unplanned follow-ups

SECONDARY OUTCOMES:
Adherence to therapy | 6 months
  Compliance data from the device
Therapy Acceptance | 6 months
  Number of withdrawals and drop out from the therapy
Apnea Hypopnea Index (AHI) | 6 months
  AHI to measure the treatment efficacy
Leak | 6 months
  Total system leak from the device
Side effects and symptoms reported | 6 months
  Any side effects and symptoms reported with the therapy
Self-reported satisfaction | 6 months
  Self-reported satisfaction via treatment questionnaires
Patient sleeping environment temperature and humidity | 6 months
  The temperature and humidity of the patient's environment as measured by a humidity logger

CONTACTS AND LOCATIONS:
Overall Officials: Sara Parsons, Chief Clinical Physiologist, Principal Investigator — Lung Function and Sleep Unit, St George's Hospital
Locations (1):
- Lung Function and Sleep Unit, St George's Hospital, London, United Kingdom